CLINICAL TRIAL: NCT07059793
Title: Post-Market Clinical Follow-up Study of Edwards Lifesciences MITRIS RESILIA Mitral Valve in Chinese Population
Brief Title: MITRIS China Post Market Clinical Follow-up (PMCF) Study
Acronym: MITRIS China
Status: Recruiting | Type: Observational
Sponsor: Edwards Lifesciences (Industry)
Collaborators: Edwards (Shanghai) Medical Products Co. Ltd. (Unknown); Kun Tuo Medical Research and Development (Beijing) Co. Ltd. (Unknown); Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-14
Record Dates: First submitted 2025-06-13; First posted 2025-07-11 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Mitral Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- MITRIS RESILIA Mitral Valve: Subjects who received the MITRIS RESILIA Mitral Valve, Model 11400M
  Interventions: Device: MITRIS RESILIA Mitral Valve

INTERVENTIONS:
Device: MITRIS RESILIA Mitral Valve — Surgical replacement of native or prosthetic mitral valve.

SUMMARY:
Collect clinical outcomes on acute and long-term safety and performance of the MITRIS RESILIA Mitral Valve, Model 11400M, in subjects requiring replacement of their native or prosthetic mitral valve with or without concomitant procedures.

DETAILED DESCRIPTION:
The trial is a Multicenter, prospective, single-arm, post-market study designed to collect clinical outcomes in up to 250 Subjects who have received the MITRIS RESILIA Mitral Valve, Model 11400M.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older at the time of informed consent
2. Has a dysfunctional native or prosthetic mitral valve and requires mitral valve replacement surgery
3. Provide signed written informed consent prior to the study participation
4. Willingness to follow protocol requirements

Exclusion Criteria:

1. Active endocarditis 3 months prior to the procedure
2. Stage 4 renal disease or requiring dialysis (eGFR < 30 is excluded)
3. Less than 2-year life expectancy due to non-cardiovascular life-threatening disease
4. High predicted risk of mortality prior to procedure - STS Predicted Risk of Mortality (PROM) > 8 or Surgeon estimated risk of mortality of > 8 (STS PROM risk calculation score must be used for patients undergoing Isolated Mitral Valve Replacement (MVR) or MVR+ Coronary Artery Bypass Grafting (CABG). Surgeon estimated risk of mortality may only be used for patients who do not qualify for evaluation against those surgical models.)
5. Participating in a drug or device study that has not reached its primary endpoint. Note: Participation in national registries is not an exclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects from China who meet all the study inclusion criteria and none of the study exclusion criteria who undergo a mitral valve replacement with the Model 11400M heart valve and voluntary sign a consent form to agree to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-07-08 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2038-12 (Estimated)

PRIMARY OUTCOMES:
Primary Safety outcome - Kaplan Meier (KM) rate of valve related death or reintervention | 1 year
  Freedom from valve related death or valve related reintervention at 1 year as determined by the CEC.
Primary Performance outcome - Hemodynamics by echocardiography - Subject's Average Mean Gradient Measurements | 1 year
  Mean gradient is the average flow of blood through the mitral valve measured in millimeters of mercury. Gradients are evaluated by echocardiography over time. In general, a higher value is considered worse, and a lower value is considered better, but the value is dependent on the size and type of valve.
Primary Performance outcome - Hemodynamics by echocardiography - Subject's Average Peak Gradients Measurements | 1 year
  Peak gradient is the maximum value measured of flow of blood through the mitral valve as measured in millimeters of mercury. Gradients are evaluated by echocardiography over time. In general, a higher value is considered worse, and a lower value is considered better, but the value is dependent on the size and type of valve.
Primary Performance outcome - Hemodynamics by echocardiography - Subject's Amount of Transvalvular regurgitation | 1 year
  Transvalvular leak is where a heart valve doesn't close properly, allowing blood to flow backward through the valve itself.
  Transvalvular leak is evaluated by echocardiography over time. It is assessed on a scale from minimum of 0 to maximum of 4, where 0 = no leak, 1 = a trace leak, 2 = a mild leak, 3 = a moderate leak, and 4 = a severe leak. Higher numbers on the scale show a worsening outcome.
Primary Performance outcome - Hemodynamics by echocardiography - Subject's Amount of Paravalvular leak | 1 year
  Paravalvular leak refers to blood flowing through a channel between the implanted artificial valve and the cardiac tissue as a result of inappropriate sealing.
  Paravalvular leak is evaluated by echocardiography over time. It is assessed on a scale from minimum of 0 to maximum of 4, where 0 = no leak, 1 = a trace leak, 2 = a mild leak, 3 = a moderate leak, and 4 = a severe leak. Higher numbers on the scale show a worsening outcome.

SECONDARY OUTCOMES:
Performance outcome - Hemodynamics by echocardiography Subject's Average Mean Gradient Measurements | 10 years
  Mean gradient is the average flow of blood through the mitral valve measured in millimeters of mercury. Gradients are evaluated by echocardiography over time. In general, a higher value is considered worse, and a lower value is considered better, but the value is dependent on the size and type of valve.
Performance outcome - Hemodynamics by echocardiography - Subject's Average Peak Gradients Measurements | 10 years
  Peak gradient is the maximum value measured of flow of blood through the mitral valve as measured in millimeters of mercury. Gradients are evaluated by echocardiography over time. In general, a higher value is considered worse, and a lower value is considered better, but the value is dependent on the size and type of valve.
Performance outcome - Hemodynamics by echocardiography - Subject's Amount of Transvalvular regurgitation | 10 years
  Transvalvular leak is where a heart valve doesn't close properly, allowing blood to flow backward through the valve itself.
  Transvalvular leak is evaluated by echocardiography over time. It is assessed on a scale from minimum of 0 to maximum of 4, where 0 = no leak, 1 = a trace leak, 2 = a mild leak, 3 = a moderate leak, and 4 = a severe leak. Higher numbers on the scale show a worsening outcome.
Performance outcome - Hemodynamics by echocardiography - Subject's Amount of Paravalvular leak | 10 years
  Paravalvular leak refers to blood flowing through a channel between the implanted artificial valve and the cardiac tissue as a result of inappropriate sealing.
  Paravalvular leak is evaluated by echocardiography over time. It is assessed on a scale from minimum of 0 to maximum of 4, where 0 = no leak, 1 = a trace leak, 2 = a mild leak, 3 = a moderate leak, and 4 = a severe leak. Higher numbers on the scale show a worsening outcome.
Adverse Events | 10 years
  Linearized rates of following key events will be presented in early (≤30 days) and late (>30 days) post-operative period. The outcomes will be adjudicated by Clinical Events Committee (CEC) up to 1 year and site-reported outcomes will be presented after completion of 1 year follow-up.
  * Thromboembolism (Stroke, Transient Ischemia Attack (TIA), Non- Cerebral)
  * Valve thrombosis
  * Major bleeding
  * Nonstructural Valve Dysfunction (NSVD)
  * Structural Valve Deterioration (SVD)
  * Endocarditis
  * Valve related reintervention
  * Death
New York Heart Association (NYHA) Classification | 10 years
  Functional improvement from baseline for NYHA Class (all follow-up time points)
  The New York Heart Association (NYHA) functional classification system relates symptoms to everyday activities and the patient's quality of life.
  Class I. No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, dyspnea (shortness of breath).
  Class II. Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea (shortness of breath).
  Class III. Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, or dyspnea.
  Class IV. Unable to carry on any physical activity without discomfort. Symptoms of heart failure at rest. If any physical activity is undertaken, discomfort increases.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Feng, Professor, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (13):
- China (13):
  - Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Fuwai Hospital, CAMS & PUMC, Beijing, Beijing Municipality
  - Xiamen Cardiovascular Hospital Xiamen University, Xiamen, Fujian
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Fuwai Central China Cardiovascular Hospital, Zhengzhou, Henan
  - Wuhan Asia Heart Hospital, Wuhan, Hubei
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Nanjing First Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of XI'an Jiaotong University, Xi'an, Shaanxi
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Ningbo Medical Center Lihuili Hospital, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: No